CLINICAL TRIAL: NCT02087501
Title: A Prospective Open-label Non-randomized Pivotal Study to Evaluate the Safety and Performance of the Horizon™ Abdominal Aortic Aneurysm (AAA) Stent Graft System
Brief Title: HORIZON CE Pivotal Study to Treat Abdominal Aortic Aneurysm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endospan Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP003.00
Record Dates: First submitted 2014-03-10; First posted 2014-03-14 (Estimated); Results first posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2022-02

CONDITIONS: Infrarenal Abdominal Aortic Aneurysms; Aortoiliac Aneurysms
Keywords: Abdominal Aortic Aneurysm; AAA; Abdominal Aortoiliac Aneurysm; Endovascular Aortic Repair; EVAR
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HORIZON AAA Stent Graft (Other): All patients will received the HORIZON AAA Stent Graft
  Interventions: Device: Horizon™ Abdominal Aortic Aneurysm Stent Graft System

INTERVENTIONS:
Device: Horizon™ Abdominal Aortic Aneurysm Stent Graft System — All patient eligible to undergo stent implantation will receive the Horizon™ Abdominal Aortic Aneurysm Stent Graft System and its designated Delivery System.

SUMMARY:
Clinical Investigation Design A prospective, open-label, non-randomized, interventional clinical study, sponsored by Endospan Ltd. Patients will be followed-up for five years.

Investigational Device The Horizon™ Abdominal Aortic Aneurysm Stent Graft System and its designated Delivery System.

Purpose The purpose of the study is to evaluate the safety and performance of the Horizon™ AAA Stent Graft System for the treatment of infrarenal abdominal aortic and/or aortoiliac aneurysms. The results of this study will be used as supportive data for CE Marking submission in the European Union (EU).

Objectives The primary objectives of the study are to evaluate the safety and performance of the Horizon™ AAA Stent graft System.

Primary End Points Safety endpoints include proportion of patients free from device related Major Adverse Events (MAEs) within 1 month of the endovascular procedure. Performance endpoints include successful delivery and deployment of the device; and absence of the following at 1 month follow-up: aneurysm growth ≥5mm, type I or III endoleaks, stent graft occlusion, conversion to open surgery, rupture and stent graft migration.

Subject population Thirty (30) patients having infrarenal abdominal aortic and/or aortoiliac aneurysms, having Iliac/femoral access vessel morphology that is compatible with vascular access techniques and devices.

Treatment All patients will be treated by implantation of the Horizon™ Abdominal Aortic Aneurysm Stent graft System.

DETAILED DESCRIPTION:
Possible benefits:

It is believed that the Horizon™ AAA Stent Graft System implantation may offer a number of benefits over conventional and recently developed treatment options for patients suffering from AAA. These other treatment modalities include open surgery and the more recently evolved EVAR.

The Horizon™ AAA Stent graft System has a low profile of 14Fr and is implanted through a percutaneous approach. The modular bottom-up construction requires a single-sided femoral access and there is no need for cannulation of the contralateral limb, a requirement present in the majority of commercially available devices. These features are anticipated to result in a simplified procedure with less surgical trauma, shorter procedure time, lower levels of radiation exposure and shorter hospitalization periods. Moreover, the device is flexible enough to reach also tortuous anatomies and its fixation elements reduce the concern of migration and type I endoleaks.

As such, it is believed that the Horizon™ AAA Stent graft System may have potential clinical advantages and may exhibit benefits over commercially available stent-grafts.

Hypothesis:

In this clinical study safety and performance primary endpoints are compared between HORIZON™ and those reported for the Lifeline Registry of Endovascular Aneurysm Repair (Control).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female age ≥ 18.
2. Presence of at least one of the following:

   i. Abdominal aortic aneurysm ≥ 5.0cm in diameter (perpendicular to the line of flow).

   ii. Abdominal aortic aneurysm 4.5-5.5cm in diameter which increased in size - ≥ 0.5cm over 6 months or 1.0cm over one year.

   iii. Abdominal aortic aneurysm >50% larger than the normal aortic diameter.
3. Patient is considered an appropriate candidate for an elective surgery, as evaluated by Physical Status Classification System I, II or III (American Society of Anesthesiologists).
4. Femoral artery diameter of ≥6mm, documented by CTA or MRA that allows endovascular access to the aneurismal site with a 14 Fr delivery catheter.
5. Access vessels morphology suitable for endovascular repair in terms of tortuosity, calcification and angulation, documented by CTA or MRA.
6. To be eligible to receive the Horizon having the following characteristics, as demonstrated on CTA or MRA imaging:

I. Infrarenal aortic diameter of 18-28 mm II. Aortic length (lower renal artery to lowest point of aortic bifurcation) of 115-150 mm III. Iliac artery diameter of 10-19 mm IV. Proximal aortic neck length ≥ 15 mm V. Proximal aortic neck angulation ≤ 60° VI. Diameter measured 20mm above aortic bifurcation floor should be ≥ 20mm VII. Aortic bifurcation angulation of ≥ 70°. 7. Patient understands and is voluntarily willing to participate as evidenced by personally signing the Informed Consent document.

Exclusion Criteria:

1. If female and of childbearing potential , patients who are:

   1. pregnant (as determined by a positive pregnancy test performed between 10 to 5 days before implantation date), or
   2. intend to become pregnant during the study period, or
   3. do not accept to use adequate double barrier contraception methods for the entire study duration to avoid pregnancy
2. Life expectancy of less than 1 year.
3. Any medical condition that, according to the investigator's decision, might expose the patient to increased risk by the investigational device or procedure.
4. Patient is in need for an emergent surgery for a ruptured aneurysm.
5. Patient with an increased risk for aneurysm rupture, such as, saccular aneurysm, aneurysm with isolated wall protrusion and penetrating ulcers of the aorta.
6. A dissecting, acutely ruptured, or leaking aneurysm, or an acute vascular injury due to trauma.
7. Presence of thrombus or atheroma in proximal aortic neck covering >50% of the endoluminal surface.
8. Presence of diffuse atherosclerotic disease in either common iliac artery that reduces the iliac artery diameter to <6mm.
9. Congenital vascular disease in which the placement of the stent graft will cause occlusion of major arterial flow.
10. Aneurysm with any of the following characteristics: suprarenal, isolated ilio-femoral, mycotic, inflammatory or para-anastomotic pseudoaneurysm.
11. Patient has an untreated thoracic aneurysm > 5.5 cm in diameter.
12. Patient has an aneurysm that involves the part of the aorta at the ostia of the renal arteries.
13. Patient has a reversed conical neck defined as a > 4mm distal increase over a 10 mm length.
14. Patient has ectatic iliac arteries requiring bilateral exclusion of hypogastric blood flow.
15. Patient whose arterial access site is not anticipated to accommodate the 14 Fr diameter of the Horizon™ Delivery System, due to size, tortuosity or hostile groins (scarring, obesity, or previous failed puncture).
16. Patient underwent major surgery or interventional procedure in the last three months.
17. Patient is suffering from unstable angina.
18. Patient has had a myocardial infarction (MI) or cerebral vascular accident (CVA) within 3 months prior to the planned implantation.
19. Patient has a known hypersensitivity or contraindication to anticoagulants, antiplatelets, or contrast media, which is not amenable to pre-treatment.
20. Contraindication to undergoing angiography.
21. Patients with known hypersensitivity or allergy to device materials - Nitinol and Polyester.
22. Morbid obesity or other clinical conditions that severely inhibit x-ray visualization of the aorta.
23. Connective tissue disease (e.g., Marfan's or Ehler's-Danlos syndromes).
24. Patient has a history of bleeding diathesis or coagulopathy.
25. Active systemic infection at the time of the index procedure documented by either one of the following: pain, fever, drainage, positive culture and/or leukocytosis (WBC > 11,000 mm3).
26. Acute renal failure documented by either one of the following: Creatinine > 2.00 mg/dl or > 182 pmol/L; patient on dialysis.
27. Any other medical, social, or psychological issues that in the opinion of the investigator preclude them from receiving this treatment, or the procedures and evaluations pre- and post- treatment.
28. Active participation in another research study involving an investigational device or new drug.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2021-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- Italy (3):
  - Nuovo Ospedale Civile S. Agostino Estense - Chirurgia vascolare, Modena
  - Azienda Ospedaliera Arcispedale S. Maria Nuova, Reggio Emilia
  - Azienda Ospedaliera Ordine Mauriziano di Torino, Torino
- Catharina Ziekenhuis Eindhoven - department of vascula surgery, Eindhoven, Netherlands
- Serbia (2):
  - Clinical Center of Serbia, Clinic for Vascular Surgery, Belgrade
  - Institute for Cardiovascular Diseases Dedinje, Belgrade
- Zurich University Hospital- Klinik für Herz- und Gefässchirurgie, Zurich, Switzerland

REFERENCES:
- [Derived] Hofmann M, Pecoraro F, Planer D, Pfammatter T, Puippe G, Bettex D, Veith FJ, Lachat M, Chaykovska L; FIM and PIVOTAL trialists. Early outcomes with a single-sided access endovascular stent. J Vasc Surg. 2018 Jul;68(1):83-90.e2. doi: 10.1016/j.jvs.2017.11.069. Epub 2018 Mar 27. PMID 29602473

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study population included 30 patients enrolled in Hospitals, enrollment period lasted 1 year.
Pre-assignment Details: There were no events occurring after patient enrollment and before assignment of the single arm foreseen by the study protocol
Groups:
- HORIZON AAA Stent Graft System: All eligible patients received the HORIZON AAA (Abdominal Aortic Aneurysm) Stent Graft System.
Period: Overall Study
Arm/Group | HORIZON AAA Stent Graft System
Started | 30
Completed | 20
Not Completed | 10
Not completed — Death | 7
Not completed — Open repair of aneurysm | 1
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Groups:
- HORIZON AAA Stent Graft: All eligible patients received the HORIZON AAA (Abdominal Aortic Aneurysm) Stent Graft System.
Arm/Group | HORIZON AAA Stent Graft
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 2
  Italy | 12
  Serbia | 11
  Switzerland | 5

OUTCOME MEASURES:

1. Primary Outcome: Safety Endpoint: Major Adverse Events (MAEs)
Description: Safety endpoint includes proportion of patients free from MAEs within 1 month post implantation, as adjudicated by an independent clinical events committee (CEC).
Time Frame: 1 month post implantation
Population: The safety analysis population consisted of all subjects for whom the implantation procedure was initiated (i.e. date of implantation was not missing).
  Out of the 30 subjects in the safety analysis set, none had Major Adverse Events (MAEs) within 1 month, and therefore the sample proportion of subjects having MAE's within 1 month is 0%. The 95% confidence interval is [0%, 11.6%], meaning that we are 95% confident that the proportion of subjects having MAE's within 1 month is lower than 11.6%.
Measure: Count of Participants; unit: Participants
Arm/Group | HORIZON AAA Stent Graft
Number analyzed (Participants) | 30
Participants | 30
Statistical Analysis 1: Comparison: HORIZON AAA Stent Graft; Test type: Other; Sample proportion = 0, 95% CI 2-sided [0 to 11.6] — The CI is calculated based on Clopper-Pearson method
Statistical Analysis 2: Comparison: HORIZON AAA Stent Graft; Test type: Other; Sample proportion = 0, 95% CI 2-sided [0 to 11.6]

2. Primary Outcome: Performance Endpoint
Description: Performance endpoints will assess the rate of successful aneurysm treatment at 1 month, defined as:
  * Successful delivery and deployment of the device.
  * Absence of the following, as determined by an independent core-lab: aneurysm growth ≥5mm, type I or III endoleaks, stent graft occlusion, conversion to open surgery, rupture and clinically significant stent graft migration.
Time Frame: 1 month post implant
Population: All subjects for whom the implantation procedure was initiated and for whom there were no major entry violations likely to affect outcome
Measure: Count of Participants; unit: Participants
Arm/Group | HORIZON AAA Stent Graft System
Number analyzed (Participants) | 30
Participants | 30
Statistical Analysis 1: Comparison: HORIZON AAA Stent Graft System; Test type: Other; Sample proportion = 100, 95% CI 2-sided [88.4 to 100] — CI is calculated based on Clopper-Pearson method

3. Secondary Outcome: MAEs
Description: Proportion of patients free from MAEs at 1 month through 5 years post implantation.
Time Frame: 1 month - 5 years post implantation
Population: All patients for whom the implantation procedure was initiated and for whom there was no major entry violation
Measure: Count of Participants; unit: Participants
Arm/Group | HORIZON AAA Stent Graft System
Number analyzed (Participants) | 30
Participants | 24
Statistical Analysis 1: Comparison: HORIZON AAA Stent Graft System; Test type: Other; Sample proportion = 80, 95% CI 2-sided [61 to 92]

4. Secondary Outcome: Mortality
Description: All-cause mortality and aneurysm-related mortality at 12 months, Kaplan-Meier survival analysis.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage free from mortality
Arm/Group | HORIZON AAA Stent Graft System
Number analyzed (Participants) | 30
percentage free from mortality | 93.3 [75.9 to 98.3]

5. Secondary Outcome: Secondary Performance Endpoint
Description: Absence of all of the following at 1 year: aneurysm growth ≥5mm, type I or III endoleaks, stent graft occlusion, conversion to open surgery, rupture and stent graft migration.
Time Frame: 12 months post implantation
Measure: Count of Participants; unit: Participants
Groups:
- HORIZON AAA Stent Graft System: All eligible patients received the HORIZON AAA (Abdominal Aortic Aneurysm) Stent Graft System. Unrelated to the aneurysm procedure deaths were excluded
Arm/Group | HORIZON AAA Stent Graft System
Number analyzed (Participants) | 28
Participants | 28

ADVERSE EVENTS:
Time Frame: For each patient, adverse events were collected for 5 years after implantation of the device.
Description: The definitions of AE and SAE follow the standard ISO14155. MAEs (used for the assessment of endpoints) are defined as: all-cause mortality, myocardial infarction, renal failure (excludes renal insufficiency), respiratory failure (excludes chronic obstructive pulmonary disease or polmunary complications), paraplegia (excludes paraparesis), stroke (excludes transient ischemic attack), bowel ischemia and procedural blood loss ≥ 1000ml.
Arm/Group | HORIZON AAA Stent Graft
All-Cause Mortality (participants affected / at risk) | 7/30
Serious Adverse Events (participants affected / at risk) | 19/30
Other Adverse Events (participants affected / at risk) | 18/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HORIZON AAA Stent Graft (N=30)
Coronary artery disease (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 3 (3)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Stent-graft endoleak (General disorders) | 2 (2)
Sudden cardiac death (General disorders) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1)
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lip and /or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Coronary artery bypass and aortic valve replacement (Surgical and medical procedures) | 1 (1)
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 (1)
Aneurysm (Vascular disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HORIZON AAA Stent Graft (N=30)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diaphragmatic hernia (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chronic fatigue syndrome (General disorders) | 1 (1)
Pirexia (General disorders) | 4 (4)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (2)
Renal cyst (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Renal infarct (Renal and urinary disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Intermittent claudication (Vascular disorders) | 1 (1)
Vasospasm (Vascular disorders) | 1 (1)
Stent-graft endoleak (General disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No